CLINICAL TRIAL: NCT00946621
Title: A Relative Bioavailability Study of Ramipril 10 mg Capsules Under Non-Fasting Conditions
Brief Title: To Demonstrate the Relative Bioavailability Study of Ramipril 10 mg Capsules Under Non-Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sandoz (Industry)
Responsible Party: Eric Mittleberg, Ph.D, VP of Product Development, Sandoz Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: B043724
Record Dates: First submitted 2009-07-24; First posted 2009-07-27 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2009-07

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Ramipril

ARMS (2):
- 1 (Experimental): Ramipril 10 mg Capsule (Sandoz)
  Interventions: Drug: Ramipril 10 mg Capsule (Sandoz)
- 2 (Active Comparator): Altace (Ramipril) 10 mg Capsule (Aventis Pharmaceutical)
  Interventions: Drug: Altace (Ramipril) 10 mg Capsule (Aventis Pharmaceutical)

INTERVENTIONS:
Drug: Ramipril 10 mg Capsule (Sandoz)
  Arms: 1
Drug: Altace (Ramipril) 10 mg Capsule (Aventis Pharmaceutical)
  Arms: 2

SUMMARY:
To demonstrate the relative bioavailability study of Ramipril 10 mg capsules under non-fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal finding on physical exam, medical history, or clinical laboratory results on screening.

Exclusion Criteria:

* Positive test results for HIV or hepatitis B or C.
* Treatment for drug or alcohol dependence.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2004-10; Primary Completion 2004-11 (Actual); Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
Bioequivalence based on AUC and Cmax | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Steven Herrmann, M.D., PhD, Principal Investigator — Cetero Research, San Antonio